CLINICAL TRIAL: NCT02336347
Title: A Phase 1, Single-center, Randomized, Double-blind, Double-dummy, 2-way Crossover Study Comparing AVP-786 With AVP-923
Brief Title: A Phase 1 Study Comparing AVP-786 With AVP-923
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Avanir Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple
Other Study IDs: 14-AVP-786-102
Record Dates: First submitted 2015-01-08; First posted 2015-01-13 (Estimated); Last update posted 2015-07-13 (Estimated); Status verified 2015-07

CONDITIONS: Healthy Volunteer
Keywords: Pharmacokinetics; Healthy Volunteers; deuterated dextromethorphan; deuterated dextromethorphan with quinidine
MeSH Terms: interventions — dextromethorphan - quinidine combination

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group 1 - Period 1 (Experimental): Twice daily dosing of AVP-786 orally for 8 days
  Interventions: Drug: AVP-786
- Group 1 - Period 2 (Active Comparator): Twice daily dosing of AVP-923 orally for 8 days
  Interventions: Drug: AVP-923
- Group 2 - Period 1 (Active Comparator): Twice daily dosing of AVP-923 orally for 8 days
  Interventions: Drug: AVP-923
- Group 2 - Period 2 (Experimental): Twice daily dosing of AVP-786 orally for 8 days
  Interventions: Drug: AVP-786

INTERVENTIONS:
Drug: AVP-786
  Other Names: deuterated (d6)-dextropmethorphan/quindine sulfate
  Arms: Group 1 - Period 1; Group 2 - Period 2
Drug: AVP-923
  Other Names: dextromethorphan/quinidine
  Arms: Group 1 - Period 2; Group 2 - Period 1

SUMMARY:
To compare pharmacokinetics (PK) of AVP-786 (deuterated [d6] dextromethorphan hydrobromide [d6-DM]/quinidine sulfate [Q]) to AVP-923 (dextromethorphan hydrobromide [DM]/Q) at steady state.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult males or females
* 18 - 60 years of age
* BMI 18 - 32 kg/m2

Exclusion Criteria:

* History or presence of significant disease
* History of substance abuse and/or alcohol abuse with the past 2 years
* Use of tobacco-containing or nicotine-containing products within 6 months
* Use of any prescription or the over-the-counter medications within 14 days

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2014-05; Primary Completion 2014-09 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
PK of d6-DM in AVP-786 compared to DM in AVP-923 | 8 days

SECONDARY OUTCOMES:
PK of metabolites | 8 days
Safety and tolerability | 8 days

CONTACTS AND LOCATIONS:
Overall Officials: Nadine Knowles, Study Director — Avanir Pharmaceuticals
Locations (1):
- Covance Dallas Clinical Research Unit, Dallas, Texas, United States